CLINICAL TRIAL: NCT00542139
Title: Evaluation of the Efficacy of Diprospan Injection to the Knee on Rehabilitation of Patients With Bilateral Knee Osteoarthritis After TKR of the Contralateral Knee.
Brief Title: Evaluation of Diprospan Injection to the Knee on Rehabilitation of Patients After TKR of the Contralateral Knee
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Leonid Kandel, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIPROSPAN- HMO-CTIL
Record Dates: First submitted 2007-10-07; First posted 2007-10-10 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2007-10

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee arthroplasty; Steroid injection; Rehabilitation
MeSH Terms: conditions — Osteoarthritis | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Betamethasone
- 2 (Active Comparator)
  Interventions: Drug: Bupivocaine

INTERVENTIONS:
Drug: Betamethasone — Intraarticular injection of 2ml Diprospan (wich contains 4mg Betamethasone sodium phosphate and 10mg Betamethasone dipropionate)
  Arms: 1
Drug: Bupivocaine — Intraarticular injection of 10ml of Bupivocaine
  Arms: 2

SUMMARY:
This study is performed to assess the influence of intraarticular injection of 2ml Diprospan (wich contains 4mg Betamethasone sodium phosphate and 10mg Betamethasone dipropionate) into osteoarthritic knee in patients who undergo a total knee replacement of their contralateral knee.

The study population will include 50 patients with bilateral knee osteoarthritis, admitted for their first knee replacement surgery. Only patients with older than 50 years with primary osteoarthritis will be included. The patients will be randomized into 2 groups. Intervention group will receive an injection of 2ml Diprospan diluted in 10 ml Bupivocaine. The control group will receive an injection of 10ml of Bupivocaine. All patients will be followed after 6 weeks and three functional rehabilitation and pain scores will be assessed (VAS pain score, Timed Up and Go Score and Functional Ambulatory Category Scale).

ELIGIBILITY:
Inclusion Criteria:

* Age older than 50
* Bilateral primary knee osteoarthritis
* Undergoing knee arthroplasty

Exclusion Criteria:

* Active infection
* Allergy to medication compounds
* Pregnancy

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Visual analogue pain score | 6 weeks

SECONDARY OUTCOMES:
Timed Up and Go Score | 6 weeks
Functional Ambulatory Category Scale | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Kandel, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel